CLINICAL TRIAL: NCT05434507
Title: Feasibility Study of Treating Tricuspid Regurgitation With K-ClipTM Transcatheter
Brief Title: Feasibility Study of Treating Tricuspid Regurgitation With K-ClipTM Transcatheter Annuloplasty System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Huihe Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH2021002
Record Dates: First submitted 2022-06-12; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- K-clipTM transcatheter annuloplasty system (Experimental)
  Interventions: Device: Transcatheter Annuloplasty

INTERVENTIONS:
Device: Transcatheter Annuloplasty — Under echocardiography guidance, the transcatheter tricuspid annuloplasty system precisely reaches the specified position in the tricuspid valve region via jugular vein and superior vena cava approach. The enlarged tricuspid annular tissue is clamped with the clamp cpart and anchor part to reduce the perimeter of tricuspid annulus, so that the area of tricuspid orifice that could not be coapted is reduced. It plays the purpose of minimally invasive treatment of tricuspid valve.

SUMMARY:
Evaluate the effectiveness and safety of the transcatheter tricuspid annuloplasty system manufactured by Shanghai Huihe Medical Technology Co., Ltd. for the treatment of patients with moderate-severe or worse tricuspid regurgitation

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60 or older, regardless of gender;
2. Patients with moderate-severe or worse tricuspid regurgitation (TR≥3+);
3. The multidisciplinary cardiac team (composed of experts in cardiovascular internal medicine and surgery, imaging, anesthesiology, etc. [No. of experts in cardiovascular surgery >=2]) considers the subjects to be at high risk for surgical operation (STS score > 6.0%) and expects that they will benefit from the transcatheter tricuspid annulus repair;
4. Patient with normal left ventricular function (LVEF≥40%);
5. The subject voluntarily participates in the clinical trial and he/she (or his/her guardian) agrees to sign the informed consent form.

Exclusion Criteria:

1. Patients with pulmonary artery systolic pressure ≥55 mmHg;
2. Patients who have a prosthetic valve or annuloplasty ring at tricuspid valve, or who underwent tricuspid valve-related treatment procedure in the past;
3. Evidence of lumps, thrombus or vegetation in the heart, jugular vein, or superior vena cava;
4. Patients with moderate or worse aortic valve stenosis, mitral stenosis, aortic regurgitation or mitral regurgitation;
5. Patients with severe uncontrolled hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg);
6. Received PCI less than 1 month ago;
7. MI happened or UAP was found less than 1 month ago;
8. CVA occurred less than 3 months ago;
9. Patients with comorbid active endocarditis or active RHD;
10. Patients with coagulation disorder, hypercoagulable state or anemia (HGB < 90 g/L);
11. Patients with acute infection or other severe infections;
12. Patients with active peptic ulcer or active gastrointestinal bleeding;
13. Patients with severe end-stage diseases (e.g., malignant tumors, severe pulmonary diseases, hepatic diseases, renal failure) whose life expectancy is less than 1 year;
14. Patients with known allergies or contraindications to the raw materials of trial product or the drugs (e.g., antiplatelet drugs, anticoagulant drugs);
15. People who are addicted to alcohol, drugs or narcotics;
16. Patients with cognitive impairment who cannot cooperate with the study or follow-up;
17. Those with a history of epilepsy or mental illness;
18. Participated in any other clinical trials (except for registry studies) less than 30 days before the signing the informed consent form;
19. Other situations that the investigator considers inappropriate for participation in this clinical trial.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Success rate 1year after operation | 1-year after operation
Success rate of operation | intra-procedure
Success rate of device implantation | intra-procedure
Change in echocardiographic parameters | 30 days, 6 Months, 12 Months, annual for five years
  Tricuspid annulus perimeter（mm）
Change in echocardiographic parameters | 30 days, 6 Months, 12 Months, annual for five years
  Tricuspid annulus area(mm2)
Change of Tricuspid Regurgitation Grade | 30 days, 6 Months, 12 Months, annual for five years
  Number of patients with reduction in TR from baseline
NYHA Functional Class | 30 days, 6 Months, 12 Months, annual for five years
  Number of patients with improvement in NYHA class
6 minutes walk distance | 1 month, 6 months,12 Months
  Increase in distance (m) from baseline
Kansas City Cardiomyopathy Questionnaire | 30 days, 6 Months, 12 Months
  Number of points of improvement in health status as measured by Kansas City Cardiomyopathy Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Huihe Healthcare Tecnology Co.,Ltd., Shanghai, Shanghai Municipality, China